CLINICAL TRIAL: NCT06518707
Title: Impact of Intraoperative Diaphragmatic Neuromodulation on Postoperative Complications in Neurosurgical Patients: A Prospective, Randomized Controlled Study
Brief Title: Intraoperative Diaphragmatic Neuromodulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Zhonghua Shi, MD, PhD, Deputy president of the department ICU, Beijing Sanbo Brain Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dia-the-Brain
Record Dates: First submitted 2024-06-18; First posted 2024-07-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Neurosurgery; Phrenic Nerve Stimulation; Postoperative Delirium
Keywords: Phrenic nerve stimulation; Postoperative delirium; Postoperative pulmonary complications
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: The intervention groups include two groups: each group will receive phrenic nerve stimulation under different degrees of neuromuscular blockade, i.e., the TOF 0 group and the TOF 1-2 group.
Who Masked: Participant, Outcomes Assessor
Masking Description: During the study period, the investigator will set the intensity of the phrenic nerve stimulation, so the investigator will not be masked. However, patients who are enrolled in this study and assessors who assess the clinical outcomes will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): No intervention will be performed; all protocols during surgery will follow the clinical routine.
- PNS + TOF 0 (Experimental): Patients in this group will receive PNS during surgery, with the train-of-four (TOF) maintained at a level of 0. Additionally, to ensure complete blockade of the neuromuscular system, the Post-Tetanic Count (PTC) will be monitored and maintained at less than or equal to 3 simultaneously.
  Interventions: Other: Phrenic nerve stimulation
- PNS + TOF 1-2 (Experimental): Patients in this group will receive PNS during surgery, and the TOF will be maintained at levels 1-2. In this group, the neuromuscular junction will not be fully blocked.
  Interventions: Other: Phrenic nerve stimulation

INTERVENTIONS:
Other: Phrenic nerve stimulation — A commercial phrenic nerve stimulation equipment will be used during surgery. Phrenic nerve stimulation intensity will be determined before surgery, ensuring significant diaphragm contraction under stimulation. The use of an electric knife will be avoided during surgery. Tidal volume, airway pressure, and vital signs will be monitored continuously.
  Arms: PNS + TOF 0; PNS + TOF 1-2

SUMMARY:
This prospective, single-center, randomized controlled clinical trial aims to investigate the impact of intraoperative phrenic nerve stimulation (i.e., diaphragmatic neuromodulation) on postoperative complications in neurosurgical patients. The primary objective is to assess the effect on postoperative brain injury, including the development of delirium and changes in biomarkers. Additionally, the incidence of postoperative pulmonary complications will be investigated.

DETAILED DESCRIPTION:
【Background】Postoperative complications, such as delirium and pulmonary complications, commonly occur in patients undergoing craniotomy. In preclinical studies, phrenic nerve stimulation (i.e., diaphragmatic neuromodulation) has been reported to effectively mitigate brain injury and pulmonary complications. However, its intraoperative administration and its impact on postoperative complications in this population are largely unknown.

【Method】In this prospective, single-center, randomized controlled clinical trial, patients receiving elective craniotomy will be screened. Eligible patients will be randomly divided into three groups: 1) Control group (without any interventions); 2) Intraoperative phrenic nerve stimulation (PNS) without total neuromuscular blockade (Train-of-Four (TOF) = 0); 3) Intraoperative PNS with partial neuromuscular blockade (TOF in the range of 1-2). Diaphragm ultrasound will be performed to assess diaphragm function before surgery and at 24 hours and 48 hours after surgery, respectively. Postoperative delirium will be assessed daily using the 3D-CAM and CAM-ICU within 3 days. Plasma biomarkers of brain injury will also be tested at baseline, 24 hours, and 48 hours after surgery. Pulmonary complications will be diagnosed by three independent clinicians based on laboratory tests, imaging, and clinical signs.

【Aims and Hypothesis】The primary aims are to investigate the impact of intraoperative diaphragmatic neuromodulation on brain injury, including the occurrence of delirium and changes in biomarkers. The secondary aims are the incidence of postoperative pulmonary complications and other clinical outcomes. We hypothesize that intraoperative diaphragmatic neuromodulation could reduce brain injury induced by craniotomy, as well as the incidence of postoperative delirium and pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Body mass index ≤ 30 kg/㎡;
* American Society of Anesthesiologists Classification: I-II level;
* Patients who undergo elective supratentorial tumor resection surgery;
* Mechanical ventilation during operation ≥ 4h;
* Signed informed consent form;

Exclusion Criteria:

* With known respiratory diseases, such as chronic obstructive pulmonary disease, obstructive sleep apnea, asthma, etc.;
* History of respiratory infection within 6 months before surgery;
* Received invasive or non-invasive mechanical ventilation within 6 months;
* Contraindications to extracorporeal diaphragmatic pacemakers, such as pneumothorax, active pulmonary tuberculosis, and wearing a cardiac pacemaker;
* Diagnosis with neuromuscular dysfunction diseases such as Guillain-Barre syndrome, myasthenia gravis, muscle atrophy, etc.;
* Pregnant or lactating patients;
* Preoperative cognitive impairment, consciousness disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium | Within 3 days after surgery
  The incidence of delirium is documented using validated delirium scores, determined by either a positive result from the 3-minute diagnostic interview for the Confusion Assessment Method (3D-CAM) scoring sheet, the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU), or both

SECONDARY OUTCOMES:
Postoperative pulmonary complications | Within 7 days after surgery
  Postoperative pulmonary complications may include respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, acute respiratory distress syndrome, aspiration pneumonia, pulmonary embolism, pulmonary edema, and aggravation of existing lung diseases.
Post operative diaphragm dysfunction | Before the surgery and within 24 hours and 48 hours after surgery.
  The patient is placed in a supine position, with a high-frequency linear array probe positioned between the right axillary midline and the 8th to 10th ribs. The probe is rotated to align parallel to the intercostal space. When two parallel high-echo lines appear, the diaphragm is identified between them. The sampling line is placed in the diaphragm movement area, and once the image stabilizes, it is converted to an M-mode ultrasound. The thickness of the inspiratory and expiratory diaphragmatic muscles is measured separately, and the maximum value is obtained by repeating the measurements three times. Diaphragm dysfunction is defined as a fraction of diaphragm thickening less than 20%.
Length of stay in Intensive Care Unit (ICU) | The time from ICU admission to transfer to the ward or death, whichever occurred first, was assessed for up to 180 days.
  The time between the patient's admission to the ICU and the patient's discharge from the ICU is referred to as the length of stay in the ICU.
Length of hospital stay | The period from hospital admission to discharge or death, whichever occurred first, was assessed for up to 180 days.
  The time between the patient's admission to the hospital and the patient's discharge from the hospital is referred to as the length of stay in the hospital.
White blood cell | Before the surgery and within 24 hours and 48 hours after surgery.
  Collect preoperative and postoperative blood routine and biochemical information from patients, specifically focusing on white blood cell counts before and after surgery.
S100 calcium-binding protein B (S-100B) | Before the surgery and within 24 hours and 48 hours after surgery.
  Evaluation of serum S-100B protein levels in patients at baseline, immediate postoperative state, and 48 hours after surgery.
Glial Fibrillary acidic protein (GFAP) | Before the surgery and within 24 hours and 48 hours after surgery.
  Evaluation of serum GFAP levels in patients at baseline, immediate postoperative state, and 48 hours after surgery.
Brain-derived neurotrophic factor (BDNF) | Before the surgery and within 24 hours and 48 hours after surgery.
  Evaluation of serum BDNF levels in patients at baseline, immediate postoperative state, and 48 hours after surgery.
Neuron-specific enolase (NSE) | Before the surgery and within 24 hours and 48 hours after surgery.
  Evaluation of serum NSE levels in patients at baseline, immediate postoperative state, and 48 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Zhonghua Shi, PhD, MD, Principal Investigator — Beijing Sanbo Brain Hospital
Locations (1):
- Beijing Sanbo Brain Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No